CLINICAL TRIAL: NCT04181970
Title: Observational Study, for Quality Assessment, of Sarcoma As a Model to Improve Diagnosis and Clinical Care of Rare Tumors Through a European and Latin American Multidisciplinary NETWORK
Brief Title: Observational Study, for Quality Assessment, of Sarcoma in European and Latin American Multidisciplinary NETWORK
Acronym: (SELNET)
Status: Recruiting | Type: Observational
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Other Study IDs: SELNET (GEIS 68)
Record Dates: First submitted 2019-06-27; First posted 2019-12-02 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Soft-tissue Sarcoma; Gastrointestinal Stromal Tumors; Bone Sarcoma
MeSH Terms: conditions — Sarcoma; Gastrointestinal Stromal Tumors; Bone Neoplasms | interventions — Quality Assurance, Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Biospecimen Retention: Samples With DNA — Formalin fixed paraffin embedded tumor sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Quality assessment — There is no intervention on study subjects. A tumor review will be performed by expert centers.

SUMMARY:
Post-authorisation, multicentric, observational, retrospective and prospective study to assess quality of care of sarcoma patients in expert and non-expert centers by analysing correlation of quality items and outcomes such as relapse free survival, overall survival, percentage of amputation, etc.

Expert pathology peer review will be performed to detect differences between expert and non-expert centers as well as differences in treatment and patient prognosis.

Tumor samples of 4 types of sarcoma would also be included in translational research to detect biomarkers and produce preclinical models.

DETAILED DESCRIPTION:
Patients with an histological diagnosis of soft-tissue sarcoma, gastrointestinal stromal tumor (GIST) or bone sarcoma (all subtypes) with ≥ 18 years old are able to be included in the study.

Data registration period includes:

Retrospective part: from January 2012 until June 2019 Prospective part: from July 2019 until January 2022.

In all clinical practice guidelines, it is recommended to refer patients with suspected sarcomas to an Expert Center (EC). The pioneers in implementing EC in sarcomas have been the Scandinavian countries, where referral is mandatory. In Spain, through the Audit of the Ministry of Health, Social Affairs and Equality, 5 CSURs (Centers, Services or Reference Units). Taken together the previous information, and since the European experience in sarcoma EC and sarcoma referral policies have shown to be positive, as numerous outcome indicators favoring patients managed in EC have been reported, a European and Latin-American consortium of sarcoma centers has emerged, supported by Horizon 2020 program (Horizon 2020 Call: H2020-SC1-BHC-2018-2020) with the aim of implementing a process to facilitate the accreditation of expert centers in sarcoma as well as a network of Latin-American sarcoma centers.

A SELNET database is available for all participating countries. to register patient's clinical data: Demographic information, Type of sarcoma (Soft-tissue/Bone/GIST), Clinical presentation, Diagnosis, Treatment, and Survival and follow-up.

Quality of care will be assessed based on the analysis of different diagnostic/therapeutic items, specified in the ESMO-EURACAN clinical practice guidelines:

* Percentage of cases > 5 cm with tru-cut biopsies.
* Percentage of biopsies carried out by sarcoma teams vs not sarcoma team (in all the series and in cases > 5 cm).
* Percentage of patients with image studies at diagnosis and before surgery.
* Percentage of patients discussed in multidisciplinary teams (MDT) before treatment.
* Percentage of patients with specified histopathological grade in pathologic report.
* Percentage of affected surgical margins in first surgery.
* Percentage of re-resections in patients with affected surgical margins in first surgery.
* Co-adjuvant therapies: percentage of patients with >5 cm, G2-3 sarcoma receiving neo/adjuvant radiotherapy.
* Percentage of patients with localized GIST with adequate risk assessment (specified mitotic count (50HPF), site and size of primary tumor).
* Percentage of patients with advanced GIST with available molecular status of KIT/PDGFR before initiating systemic therapy for advanced disease.
* Percentage of patients with regular follow-up.

For the localised disease quality assessment, we'll focus on:

* Surgical margins will be correlated with: Type of biopsy, team performing diagnostic biopsy, preoperative image studies and discussion in MDT.
* Relapse-free survival will be correlated with type of biopsy, team performing diagnostic biopsy, discussion in MDT, surgical margins status, re-resection performance, co-adjuvant therapies
* Overall survival will be correlated with team performing diagnostic biopsy, discussion in MDT, surgical margins status, re-resection performance, coadjuvant therapies
* Percentage of amputation will be correlated with type of biopsy, team performing diagnostic biopsy, discussion in MDT, surgical margins status.
* Long-term side effects will be correlated with type of surgery, team performing diagnostic biopsy, discussion in MDT, surgical margins status, co-adjuvant therapies.

For advance disease quality assessment, we'll focus on:

* Progression-free survival will be correlated with discussion in MDT, type of center (expert/not)
* Overall survival will be correlated with discussion in MDT, access to clinical trials, access to second lines, surgery of metastatic disease, type of center (expert/not)

An expert pathology review will take place to diagnose sarcoma cases and evaluate the differences in diagnosis and it outcome and consequences.

Four sarcoma subtypes have been selected to analyse further with biological tissue samples.: Angiosarcoma, Desmoplastic Small Round Cell Tumor, Extraskeletal myxoid chondrosarcoma and Solitary fibrous tumors. The aims of the translational research program are: to describe prognostic factors and/ or cell signaling pathways of relevance in AS, DSRCT, EMC and SFT; to describe predictive biomarkers of first and second line agents; to study the potential mechanisms of action of first and second line agents and their role in the activation of antitumor tumor microenvironment (e.g. immune response) and to establish preclinical models on these rare subtypes of sarcoma to validate OMICs data. This will open new doors for novel hypothesis for clinical trials based on the analysis of differential gene expression, cell signaling pathways and/ or predictive biomarkers.

Progression Free Survival (PFS), objective tumor response, Overall survival (OS), and histopathological features will be correlated with OMICs data.

Samples to collect:

* Tumor blocks will be used to analyze protein fusion (by NGS), RNA expression (by RNA-Seq) and protein expression (by IHC). The tumors samples will be collected from the diagnostic time. If available, paired tumor samples will be shipped to determine the differential gene expression of post-treatment specimens.
* Prospective fresh tumor samples will be used for whole genome sequencing and to establish PDX and 3D tumor organoid-like models, at translational central laboratories (SFT: Seville; EMC: Milan; AS: Lyon; DSRCT; Sao Paulo).Moreover, fresh tumor samples could also be collected, from national associated centers, and shipped frozen to national central laboratory. Frozen tumors will be shipped in 10% DMSO - 90% FBS, which preserves quite well tumor cell viability.

All patients should sign and date the Informed Consent Form after reading the patient Information Sheet to accept participating in this study. Participating in the study is voluntary and the patient can withdraw his/her consent at any time, without giving any reason and without reducing his/her right to health care.

He/she can also withdraw the consent to use the tumor sample donated to the study without withdrawing the participation in the study (the patient's clinical data will be registered and analysed). If this happens, the tumor sample left in the central laboratory can be returned to the origin site. Any withdraw should be confirmed by signing a Revocation Form. However, the investigator should try to know the reason to withdraw consent in order to improve the study conditions.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of soft-tissue sarcoma, GIST or bone sarcoma (all subtypes) from January 2005 until Juny/September 2023.
* ≥ 18 years
* Available clinical and treatment information

Exclusion Criteria:

There is no exclusion criteria

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Soft-tissue sarcoma, Gastrointestinal stromal tumor (GIST) Bone sarcoma (all subtypes)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases with > 5 cm with tru-cut biopsies. | through study completion, an average of 3 years
  tumor should be bigger than 5cm
Percentage of biopsies carried out by sarcoma teams vs not sarcoma team | through study completion, an average of 3 years
  in all the series and in cases with > 5 cm
Percentage of patients with image studies at diagnosis and before surgery. | through study completion, an average of 3 years
  The same type of image should have been performed
Percentage of patients discussed in Multidisciplinary Team before treatment | through study completion, an average of 3 years
  multidisciplinary team includes serval departments at the same center
Percentage of patients with specified histopathological grade in pathologic report. | through study completion, an average of 3 years
  Using FNCLCC grade criteria
Percentage of affected surgical margins in first surgery | through study completion, an average of 3 years
  Using Enneking classification for determinations of surgical margins
Percentage of re-resections in patients with affected surgical margins in first surgery | through study completion, an average of 3 years
  Using Enneking classification for determinations of surgical margins
percentage of patients with >5 cm and G2-3 sarcoma receiving neo/adjuvant radiotherapy | through study completion, an average of 3 years
  Using FNCLCC grade criteria
Percentage of patients with localized GIST with adequate risk assessment | through study completion, an average of 3 years
  Classifying risk with mitotic count (50HPF), site and size of primary tumor
Percentage of patients with advanced GIST with available molecular status of KIT/PDGFR before initiating systemic therapy for advanced disease | through study completion, an average of 3 years
  Detection of KIT/PDGFR y Sanger and or NGS

SECONDARY OUTCOMES:
Surgical margins | through study completion, an average of 3 years
  using Enneking
Relapse-free survival | tthrough study completion, an average of 3 years
  days of survival from date of first line treatment until progression or death
Overall survival | through study completion, an average of 3 years
  Days from diagnosis (date of biopsy or first pathology report) until death whatever cause.
Percentage of amputation | through study completion, an average of 3 years
  Resection of any member.

CONTACTS AND LOCATIONS:
Overall Officials: Javier MARTIN-BROTO, MD, Principal Investigator — Salud de Madrid
Locations (9):
- Alexander Fleming Sa, Buenos Aires, Argentina
- A C Camargo, São Paulo, Brazil
- Hospital San Vicente de Paúl, Heredia, Costa Rica
- Centre Leon Berard, Lyon, France
- Italy (2):
  - Instituto Ortopedico Rizzoli, Bologna
  - Insituto Nazionale Di Tumore, Milan
- Instituto Nacional de Cancerología, Mexico City, Mexico
- Instituo Nacional de enfermedades Neoplásicas, Surquillo, Peru
- Fundación Jiménez Díaz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data could be shared receiving an application to the Study Main contact indicating reason and objectives.